CLINICAL TRIAL: NCT03293719
Title: Prospective, Open, Non-randomized, Non-interventional Explorative, Comparative, Uncontrolled Cohort Study for Post Market Clinical Follow-Up of the "BPK-S Integration" UC in the Variants CoCr or Ceramic as Primary Implant
Brief Title: Post-market Follow up Study of the 'BPK-S Integration' UC as Primary Implant in the Variants CoCr or Ceramic
Status: Terminated | Type: Observational
Why Stopped: Monocentric Study, Site reorganised, could no longer participate in study
Sponsor: Peter Brehm GmbH (Industry)
Collaborators: P.R.I.S.M.A.-CRO (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2017-02-BPK-S Comparison
Record Dates: First submitted 2017-09-19; First posted 2017-09-26 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee; Joint Instability; Arthritis; Joint Disease; Musculoskeletal Disease; Rheumatic Diseases
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Joint Instability; Arthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ceramic: Patients receiving BPK-S Integration UC implant made from BIOLOX delta ceramic
  Interventions: Device: BPK-S Integration UC
- CoCr: Patients receiving BPK-S Integration UC implant made from CoCr (metal)
  Interventions: Device: BPK-S Integration UC

INTERVENTIONS:
Device: BPK-S Integration UC — Primary Knee Endoprosthesis

SUMMARY:
Prospective Post-Market Clinical Follow up study according to MEDDEV 2.12/2 rev2 of the European Union. Patients receiving the primary knee implant BPK-S UC as primary implant in either variant ceramic or CoCr (metal) are eligible for the study and will be followed up for 5 years after implantation or until revision of the prosthesis, whichever occurs first. Demographic data will be collected together with data regarding safety and benefit at defined timepoints (preoperative, intraoperative and at 3 months, 1 year, 2 years and 5 years after implantation).

Patients will be divided in 2 cohorts (ceramic and metal) and stratified by age.

ELIGIBILITY:
Inclusion Criteria:

* Congenital or acquired knee joint defects/deformation
* Defects or malfunction of the knee joint
* Arthrosis (degenerative, rheumatic)
* Post-traumatic arthritis
* Symptomatic knee instability
* Reconstruction of flexibility
* Patients with metal hypersensitivity (ceramic tibia/femur)

Exclusion Criteria:

* Illnesses which can be treated without using a knee joint implant.
* Acute or chronic infections near the implantation
* Systemic diseases and metabolic disorders
* Serious osteoporosis
* Serious damage to the bone structures that impedes stable implantation of the implant components
* Diseases that impair bone growth, e.g. cancer, renal dialysis, osteopenia, etc.
* Bone tumors in the area of the implant anchoring
* Obesity or overweight of the patient
* Overload of the knee implant to be expected
* Abuse of medication, drug abuse, alcoholism or mental disease
* Pregnancy
* Lack of patient cooperation
* Sensitivity to foreign matter in the implant materials
* Patients under the age of 18
* Patients participating in another trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing primary total knee endoprosthesis with BPK-S Integration of age 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Patient relevant benefit after 5 years | 5 years
  improvement of KSS-Score by at least one category as compared to preoperative basic assessment

SECONDARY OUTCOMES:
Patient relevant benefit as measured by American Knee Society Score | 3 months, 1, 2 and 5 years
  improvement of KSS-Score as compared to preoperative basic assessment
Patient relevant benefit as measured by Knee Osteoarthritis Outcome Score | 3 months, 1, 2 and 5 years
  Improvement of KOOS as compared to preoperative basic assessment
Patient Quality of Life | 3 months, 1, 2 and 5 years
  Improvement of EQ-5D as compared to preoperative basic assessment
Implant Loosening Number | 3 months, 1, 2 and 5 years
  Number of implant loosening due to quality issues with the implant
Implant Loosening Reason | 3 months, 1, 2 and 5 years
  Reason for implant loosening due to quality issues with the implant
Revision Number | 3 months, 1, 2 and 5 years
  Number of revisions, if required
Revision Reason | 3 months, 1, 2 and 5 years
  Reason for revision, if required

CONTACTS AND LOCATIONS:
Overall Officials: Christian E. Berger, Prof., Principal Investigator — Sozialmedizinisches Zentrum Ost - Donauspital
Locations (1):
- SMZ Ost, Donauspital, Vienna, Upper Austria, Austria